CLINICAL TRIAL: NCT07345455
Title: Effect of Probiotics on Sperm Quality in Male Infertility Patients
Brief Title: Probiotics on Sperm Quality in Male Infertility Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GP001
Record Dates: First submitted 2025-05-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-01

CONDITIONS: Male Infertility; Oligozoospermia; Asthenozoospermia; Teratozoospermia; Oligoasthenoteratozoospermia
Keywords: Probiotics; Sperm Motility; Sperm DNA; Sperm Function; Oligozoospermia; Asthenozoospermia
MeSH Terms: conditions — Infertility, Male; Oligospermia; Asthenozoospermia; Teratozoospermia | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This project will collect 60 male infertility patients (mainly those with oligozoospermia and asthenozoospermia) for a period of two years and divide them into an experimental group and a control group. The experimental group was given probiotics, while the control group was given the same dosage form without probiotics (placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The control group receives a placebo identical in dosage form and appearance to the probiotic supplement, to ensure masking of participants and investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Probiotics Group (Experimental): The experimental group takes probiotics, two capsules a day, after meals.
  Interventions: Dietary Supplement: Probiotics
- Placebo Comparator: Control Group (Placebo Comparator): The control group is given the same dosage form without probiotics (placebo), two capsules a day, after meals.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — The subjects take 2 probiotic capsules after each meal daily.
  Arms: Experimental: Probiotics Group
Dietary Supplement: Placebo — The control group takes two placebo capsules (containing no probiotics) after meals daily.
  Arms: Placebo Comparator: Control Group

SUMMARY:
This randomized, placebo-controlled pilot study aims to evaluate the effects of probiotic supplementation on sperm quality in male patients diagnosed with infertility. Male infertility accounts for approximately 40% of all infertility cases and is closely related to abnormalities in sperm count, motility, and morphology. Factors such as oxidative stress, inflammation, and DNA fragmentation are known to impact sperm function and subsequent fertilization potential negatively.

Probiotics are microorganisms that confer health benefits by improving the intestinal microenvironment and regulating immunity. Emerging research suggests that probiotics may reduce oxidative stress and DNA fragmentation in men with asthenozoospermia; however, clinical data on human sperm remains limited. This study seeks to determine whether specific probiotic strains can improve sperm parameters and function in patients with unexplained oligozoospermia, asthenozoospermia, or oligoasthenoteratozoospermia.

The study will enroll 60 male participants aged 20 to 45 who meet specific inclusion criteria, including a sperm concentration of less than 50 million/mL, motility less than 40%, and normal morphology (Kruger) less than 4%. Participants will be randomly assigned to either an experimental group receiving probiotics or a control group receiving a placebo for approximately 100 days.

Semen samples will be collected and analyzed at three time points: before the intervention (Day 0), during the intervention (Day 60), and at the end of the study (Day 100). The primary objective is to assess changes in sperm concentration, motility, and morphology using the Computer-Aided Sperm Analysis (CASA) system. Secondary objectives include evaluating sperm DNA integrity using the Sperm Chromatin Structure Assay (SCSA) by flow cytometry and assessing sperm function via the acrosome reaction assay. The results of this pilot study will help determine the potential therapeutic role of probiotics in the management of male infertility.

DETAILED DESCRIPTION:
Content: Male infertility accounts for approximately 40% of infertility cases and is often characterized by abnormalities in sperm count, motility, and morphology. Factors such as oxidative stress, environmental hormones, and inflammation can lead to sperm DNA fragmentation and mitochondrial dysfunction, ultimately affecting fertilization potential. While probiotics are known to improve gut microbiome balance and regulate immunity, limited studies suggest they may also improve sperm motility and reduce DNA fragmentation in men with asthenozoospermia.

This pilot study employs a randomized, placebo-controlled design to evaluate the efficacy of probiotic supplementation in improving sperm quality. A total of 60 male participants with unexplained infertility (specifically oligozoospermia, asthenozoospermia, or oligoasthenoteratozoospermia) will be recruited. Participants will be divided into two groups: an experimental group receiving probiotics and a control group receiving a placebo.

The study duration for each participant is approximately 100 days, with semen samples collected at three distinct time points:

1. Day 0 (Start Test): Baseline sample collection.
2. Day 60 (Mid Test): Interim sample collection.
3. Day 100 (Final Test): Post-intervention sample collection.

Semen analysis will be conducted using the following methodologies:

* Sperm Concentration and Motility: Analyzed using a Computer-Aided Sperm Assay (CASA) to measure parameters including total motility, progressive motility, VAP, VCL, VSL, Straightness, and Linearity.
* Sperm DNA Integrity: Assessed via the Sperm Chromatin Structure Assay (SCSA) using flow cytometry. Sperm are treated with acridine orange; red fluorescence indicates single-stranded DNA (fragmentation), while green fluorescence indicates double-stranded DNA. Results are expressed as the DNA Fragmentation Index (DFI).

Sperm Function (Acrosome Reaction): Evaluated using Peanut Agglutinin (PNA) staining. The assay determines the percentage of sperm capable of undergoing the acrosome reaction, a necessary step for fertilization.

Inclusion Criteria

* Gender: Male.
* Age: 20 to 45 years old.
* Diagnosis: Diagnosed with unexplained oligozoospermia, asthenozoospermia, or oligoasthenoteratozoospermia.
* Semen Parameters:

  * Sperm concentration < 5×106/mL (Note: Source indicates "5x10/mL", contextually adjusted to standard unit for oligozoospermia).
  * Sperm motility < 40%.
  * Sperm morphology (Kruger strict criteria) < 4%. Exclusion Criteria

    1. History of hormonal disorders or epididymo-orchitis.
    2. Substance abuse, including drugs or excessive alcohol consumption.
    3. Diabetes mellitus.
    4. Kidney disease (defined as a doubling of creatinine levels or more).
    5. Chronic liver disease.
    6. Varicocele.
    7. Current use of medications that interfere with hormones.
    8. Occupational or environmental exposure to pesticides, heavy metals, or solvents.
    9. Intake of antioxidant supplements within the past three months.
    10. Body Mass Index (BMI) of 30 kg/m² or higher.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 20 to 45 years
* Diagnosis of unexplained oligozoospermia, asthenozoospermia, or oligoasthenoteratozoospermia
* Sperm concentration < 5 x 10^6/mL
* Sperm total motility < 40%
* Sperm morphology (Kruger strict criteria) < 4%

Exclusion Criteria:

* History of hormonal disorders or epididymo-orchitis
* Substance abuse, including drugs or excessive alcohol consumption
* Diabetes mellitus
* Kidney disease (defined as a doubling of creatinine levels or more)
* Chronic liver disease
* Varicocele
* Current use of medications that interfere with hormones
* Occupational or environmental exposure to pesticides, heavy metals, or solvents
* Intake of antioxidant supplements within the past three months
* Body Mass Index (BMI) of 30 kg/m^2 or higher

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Sperm Concentration Assessed by Computer-Aided Sperm Analysis (CASA) | Day 60, Day 100
  Sperm concentration (million/mL) will be measured using the Computer-Aided Sperm Analysis (CASA) system. The change from Baseline (Day 0) to subsequent time points will be calculated.
Change From Baseline in Total Sperm Motility Percentage Assessed by Computer-Aided Sperm Analysis (CASA) | Day 60, Day 100
  The percentage of total motile sperm will be measured using the Computer-Aided Sperm Analysis (CASA) system. The change from Baseline (Day 0) to subsequent time points will be calculated.
Change From Baseline in Percentage of Normal Sperm Morphology Assessed by Computer-Aided Sperm Analysis (CASA) | Day 60, Day 100
  The percentage of sperm with normal morphology will be measured based on Kruger strict criteria using the Computer-Aided Sperm Analysis (CASA) system. The change from Baseline (Day 0) will be calculated.

SECONDARY OUTCOMES:
Change From Baseline in Sperm DNA Fragmentation Index (DFI) Assessed by SCSA | Day 60, Day 100
  Sperm DNA integrity will be assessed using the Sperm Chromatin Structure Assay (SCSA) via flow cytometry. Sperm are stained with acridine orange. The result is expressed as the DNA Fragmentation Index (DFI), representing the ratio of red fluorescence (fragmented DNA) to total fluorescence (red + green). A lower DFI indicates better DNA integrity.
Change From Baseline in Sperm Acrosome Reaction Rate Assessed by PNA Staining | Day 60, Day 100
  Sperm function will be evaluated by the acrosome reaction assay using peanut agglutinin (PNA) staining. The percentage of sperm that have undergone the acrosome reaction (indicated by specific staining patterns observed under a fluorescence microscope) will be calculated. This measures the sperm's physiological capability to fertilize an egg.

CONTACTS AND LOCATIONS:
Locations (1):
- MacKay Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided